CLINICAL TRIAL: NCT04407364
Title: The CoMatryx Surgical Collagen Powder is a Soft Tissue Repair Product Made of 100% Type I Bovine Collagen
Brief Title: MPM Medical CoMatryx Surgical Bovine Collagen Study
Status: Active, not recruiting | Type: Observational
Sponsor: MPM Medical (Industry)
Collaborators: Texas Health Resources (Other)
Responsible Party: Sponsor
Other Study IDs: MPMCOM20
Record Dates: First submitted 2020-05-20; First posted 2020-05-29 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Surgical Wound, Healed
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Intervention Cohort: The CoMatryx surgical collagen powder is a soft tissue repair product made of 100% type I bovine collagen
  Interventions: Device: CoMatryx Surgical Bovine Collagen
- Historical Cohort: Primary and Revision total hip arthroplasty patients between 18-85 years of age
  Interventions: Device: CoMatryx Surgical Bovine Collagen

INTERVENTIONS:
Device: CoMatryx Surgical Bovine Collagen — The CoMatryx surgical collagen powder is a soft tissue repair product made of 100% type I bovine collagen
  Other Names: Interventional Cohort; Historical Cohort with no intervention

SUMMARY:
The objective of this prospective enrollment study is to collect data confirming safety, performance and clinical benefits of the CoMatryx Surgical Collagen powder at a minimum 1-year follow-up and compare it to a historical control group who did not receive the product at the time of surgery.

The primary objective is to confirm safety and clinical benefits of the product. This will be assessed by recording the rate of wound healing and incidence and frequency of wound care related complications. Relationship of complications to the product should be specified.

DETAILED DESCRIPTION:
The CoMatryx Surgical Collagen powder is a soft tissue repair product made of 100% Type I Bovine collagen. It is non-hydrolyzed and not cross-linked chemically. It is biocompatible, biodegradable and free of synthetics. The product does not have any specific storage requirements.

The CoMatryx Surgical Collagen powder provides a physiologically favorable environment to promote healing at the wound site. When administered, the powder conforms to the wound site and forms a gelatinous occlusive barrier. Along with providing 19 amino acids directly to the wound site it also occludes live nerve endings reducing pain. Treating the wound with the CoMatryx Surgical Collagen powder provides the non-hydrolyzed collagen wound surface promoting autolytic debridement. The powder is effective in all phases of wound healing and can be delivered with antibiotics in areas where there may be a cavity. This product has FDA 510(k) clearance for surgical wounds, full thickness wounds, traumatic wounds and skin tears.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects must be 18 years of age or older

  * Subject must be willing and able to sign IRB approved informed consent
  * Subject must have a BMI of 35 or higher
  * Surgical approach of only ASI (anterior supine)
  * Primary total hip arthroplasty
  * Revision total hip arthroplasty

Exclusion Criteria:

* • Subjects more than 85 years of age

  * Subjects who will be or have undergone bilateral total hip replacements
  * Subject is known to be pregnant or nursing
  * Subject is an alcohol or drug abuser
  * Subject has a psychiatric illness or cognitive deficit that will not allow for proper informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary and Revision total hip arthroplasty patients between 18-85 years of age
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
CoMatryx Surgical Bovine Collagen | This study will require following-up with patients up to 1-year post surgery. The estimated time of completion from enrollment (100 patients) to completing 1 year follow-up is 2 years.
  The primary objective is to confirm safety and performance of the study product. This will be assessed by recording the rate of healing, incidence and frequency of complications and adverse events relative to the surgical incision at 1-week, 2-week, 6-week, 6-month and 1-year follow-up. Height and Weight will be combined as BMI(kg/m^2)
CoMatryx Surgical Bovine Collagen Height and Weight | This study will require following-up with patients up to 1-year post surgery. The estimated time of completion from enrollment (100 patients) to completing 1 year follow-up is 2 years.
  Height and Weight will be combined as BMI(kg/m^2)

SECONDARY OUTCOMES:
Bovine Collagen | This study will require following-up with patients up to 1-year post surgery. The estimated time of completion from enrollment (100 patients) to completing 1 year follow-up is 2 years.
  The secondary objective is the assessment of clinical benefits by analyzing recorded subject-reported pain scores

CONTACTS AND LOCATIONS:
Overall Officials: Kwame Ennin, MD, Principal Investigator — Texas Health Physicians Group
Locations (1):
- Texas Center for Joint Replacement, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No